CLINICAL TRIAL: NCT05496803
Title: Chung Shan Medical University Hospital
Brief Title: Impact of Systematic Nursing Guidance on the Psychological Effects of Parents of Children With Cardiac Catheterization.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung Shan Medical University Hospital (Other)
Responsible Party: Sponsor-Investigator, Chung Shan Medical University Hospital, Department of pediatrics, Chung Shan Medical University
Organization: Chung Shan Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CS2-22078
Record Dates: First submitted 2022-08-03; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Educational Videos; Catheterization; Congenital Heart Disease in Children; Parental Uncertainty; Parental Anxiety

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Other): parents receiving routine education plus digital video disk before catheterization:pre-catheterization educational videos plus routine education
  Interventions: Other: routine education plus digital video disk
- control group (Other): parents receiving routine education: pre-catheterization routine education
  Interventions: Other: routine education

INTERVENTIONS:
Other: routine education plus digital video disk — Parents receiving routine education plus digital video disk before their children receiving congenital heart disease catheterization. The DVD content was the same as the routine education but was presented audio-visually, and the video was easy to understand by the general public.
  Arms: study group
Other: routine education — Parents receiving routine education before their children receiving congenital heart disease catheterization
  Arms: control group

SUMMARY:
To examine if adding educational digital video disk to routine education can reduce parental uncertainty and anxiety more if their children undergo congenital heart disease catheterization and when catheterization or post- catheterization complications occur. We want to know, compared to only routine education, if adding digital video disk could decrease parental uncertainty or anxiety more or not.

DETAILED DESCRIPTION:
Aims and objectives: To examine if adding educational digital video disk to routine education can reduce parental uncertainty and anxiety more if their children undergo congenital heart disease catheterization and when catheterization or post- catheterization complications occur.

Background: Parents experience uncertainty and anxiety when their children undergo conditions mentioned above.

Design: A randomized control-group pretest-posttest design. Methods: In a teaching hospital, 50 fathers and 50 mothers whose children (n=50) underwent first elective catheterization for congenital heart disease were randomly divided into group 1: 25 fathers and 25 mothers receiving routine education plus digital video disk before catheterization; and group 2: 25 fathers and 25 mothers receiving routine education before catheterization. Between groups, parental uncertainty and anxiety levels were compared (1) before education, (2) after education (before catheterization) and (3) on the discharge day (after catheterization). Among mothers whose children had catheterization or post- catheterization complications, the effect of watching the digital video disk on uncertainty and anxiety at discharge day was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Parents whose children underwent first elective cardiac catheterization for congenital heart disease
* Parents should have been the primary caregivers
* Parents able to communicate effectively, either orally or in writing

Exclusion Criteria:

* Parents of children with genetic disorders
* Parents of children with non-cardiac congenital anomalies
* Parents of children with diseases such as cerebral palsy, epilepsy, psychiatric diseases, and chronic lung diseases

Ages: 20 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
The change of parental uncertainty | day 1 (baseline, before education), day 1 (after education), day 2-5 (discharge day)
  The scores of parental uncertainty between "routine education" and "routine plus DVD education" groups.
  parent's perception uncertainty in illness score was used to evaluate the number scores of anxiety.
The change of parental anxiety 1 | day 1 (baseline, before education), day 1 (after education), day 2-5 (discharge day)
  The number scores of parental anxiety between "routine education" and "routine plus DVD education" groups.
  State Anxiety Inventory was used to evaluate the number scores of anxiety.
The change of parental anxiety 2 | day 1 (baseline, before education), day 1 (after education), day 2-5 (discharge day)
  The number scores of parental anxiety between "routine education" and "routine plus DVD education" groups.
  Beck Anxiety Inventory was used to evaluate the number scores of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University Hospital., Taichung, Taiwan